CLINICAL TRIAL: NCT06704711
Title: The Effect of Incremental Exercise After Caffeine Mouth Rinse on Salivary Immunoglobulin A, Lactoferrin and A-Amylase Levels
Brief Title: Caffeine Mouth Rinse on Salivary Immunoglobulin A, Lactoferrin and A-Amylase Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Cemre Didem Eyipinar, Cemre Didem EYIPINAR, University of Gaziantep
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E-87841438-100-567059
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Exercise Response
Keywords: Sportomics; Salivary immunuglobulin-a; salivary lactoferrin; salivary a-amylase; caffeine
MeSH Terms: interventions — Caffeine; Exercise

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, placebo-controlled crossover trial design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Caffeine Mouth Rinse with incremental exercise (Experimental): They will rinse a solution containing a total of 400 mg caffeine (20 mL, 2% concentration) in the mouth for 20 seconds and try to continue the exercise against increasing resistance until exhaustion. The exercise test will be performed on a bicycle ergometer (Ergometer Exercise Bike SANA 500, Germany) (where the pedaling speed is kept constant at 60 rpm, with an initial load of 50 Watts and a load increase of 25 watts per minute, gradually increasing until the participants become exhausted. To be able to determine the degree of difficulty perceived during the test and The Borg Scale will be used to end the test when the athlete reaches the point of exhaustion.
  Interventions: Dietary Supplement: Caffeine 300 MG; Combination Product: Exercise
- Placebo Rinse with incremental exercise (Placebo Comparator): They will rinse 20 mL of distilled water in the mouth for 20 s and try to continue the exercise against increasing resistance until exhaustion.The exercise test will be performed on a bicycle ergometer (Ergometer Exercise Bike SANA 500, Germany) (where the pedaling speed is kept constant at 60 rpm, with an initial load of 50 Watts and a load increase of 25 watts per minute, gradually increasing until the participants become exhausted. To be able to determine the degree of difficulty perceived during the test and The Borg Scale will be used to end the test when the athlete reaches the point of exhaustion.
  Interventions: Combination Product: Exercise; Other: Placebo
- Control Group (Experimental): Only rinse a solution containing a total of 400 caffeine (20 mL, 2% concentration) in the mouth for 20 seconds and receive no exercise treatment.
  Interventions: Dietary Supplement: Caffeine 300 MG

INTERVENTIONS:
Dietary Supplement: Caffeine 300 MG — They will rinse the solution containing a total of 400 mg of caffeine (20 mL, 2% density) in the mouth for 20 seconds and try to continue the exercise against increasing resistance until exhaustion.
  Arms: Caffeine Mouth Rinse with incremental exercise; Control Group
Combination Product: Exercise — The exercise test will be performed on a bicycle ergometer (Ergometer Exercise Bike SANA 500, Germany) (where the pedaling speed is kept constant at 60 rpm, with an initial load of 50 Watts and a load increase of 25 watts per minute, gradually increasing until the participants become exhausted. To be able to determine the degree of difficulty perceived during the test and The Borg Scale will be used to end the test when the athlete reaches the point of exhaustion.
  Arms: Caffeine Mouth Rinse with incremental exercise; Placebo Rinse with incremental exercise
Other: Placebo — They will rinse 20 mL of distilled water in their mouth for 20 seconds.
  Arms: Placebo Rinse with incremental exercise

SUMMARY:
The goal of this clinical trial is to investigate the effects of the mouth rinse form of caffeine (400 mg) on salivary lactoferrin, α-amylase and secretory immunoglobulin-a levels after incremental exercise in young amateur football players. The main questions it aims to answer are:

* Caffeine in mouth rinse form increases salivary immunoglobulin a after incremental exercise
* Caffeine in mouth rinse form increases salivary lactoferrin after incremental exercise
* Caffeine in mouth rinse form increases salivary a-amylase after incremental exercise.

This 3-session study will use a double-blind, randomized, placebo-controlled crossover experimental design. participants will complete three different treatments [caffeine (CAF), control (C) and placebo (PLA)] separated by at least 1 week. Baseline saliva samples will be collected while sitting in a chair and then:

* CAF Group: They will rinse a solution containing a total of 400 mg caffeine (20 mL, 2% concentration) in the mouth for 20 seconds and try to continue the exercise against increasing resistance until exhaustion.
* Control Group: Only rinse a solution containing a total of 400 caffeine (20 mL, 2% concentration) in the mouth for 20 seconds and receive no exercise treatment.
* Placebo Group: They will rinse 20 mL of distilled water in the mouth for 20 s and try to continue the exercise against increasing resistance until exhaustion.

Saliva samples will be collected at 6 different time points: 5 minutes before exercise (or caffeine mouth rinse) (T0-reference), immediately after caffeine mouth rinse (or immediately before exercise) (T1), 5 minutes/midway through exercise (T2), and immediately after exercise (T3), 60 minutes after the end of exercise (T4) and 120 minutes after the end of exercise (T5).All data will be statistically analyzed using SPSS 25.0 software (Chicago, IL, USA) and expressed as mean ± standard deviation. Shapiro-Wilk and Levene tests will be used to determine whether the data are normally distributed and whether the variance is homogeneous. Repeated measures ANOVA test will be used to compare group means. If there is a difference between the groups as a result of the analysis, post-hoc tests will be used to find out from which group this difference originates. In cases where the data are not normally distributed, nonparametric test methods will be used. The significance level of the tests will be accepted as p<0.05

ELIGIBILITY:
Inclusion Criteria:

* Healthy men who have not had any previous injuries, do not have a chronic disease, do not use medication, do not smoke, and have played or are playing football as an amateur.

Exclusion Criteria:

Those who have had any previous injury, have a chronic disease, use medication, or smoke.

-

Ages: 19 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-12-16 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Salivary antimicrobial proteins (Salivary a-amylase, lactoferrin and Ig-A) | From enrollment to the end of treatment at 4 weeks
  Salivary A-Amylase: Amylase functions as an antibacterial protein that inhibits bacterial growth and colonization in the oral cavity.
  Salivary Lactoferrin: Lactoferrin, one of the most abundant salivary antimicrobial proteins, exerts an antibacterial effect by retaining iron, an essential nutrient for bacterial growth, and also by directly interacting with and damaging bacterial membranes.
  Salivary Immunuglobulin-A: Salivary IgA (SIgA) contributes to mucosal immunity by preventing pathogens from adhering to the mucosal surface.

SECONDARY OUTCOMES:
Rating of Perceived Exertion | From enrollment to the end of treatment at 4 weeks
  It is defined as "felt strain" in terms of training.

IPD SHARING:
Plan to Share IPD: Yes
I want to ensure that the study reaches all researchers with the link I will receive from here.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code